CLINICAL TRIAL: NCT07056413
Title: BRILMA Block: A Regional Approach to Pain Management in Breast-Conserving Surgery
Brief Title: BRILMA Block in Breast-Conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nukhet Sivrikoz, Attending Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/676
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
Keywords: BRILMA block; breast-conserving surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B: BRILMA block (Experimental): 20 ml 0.25 % bupivacaine was injected into the fascial plane between the serratus anterior muscle and the external intercostal muscle at T4 level.
  Interventions: Procedure: BRILMA block
- Group C: Control (Other): Standard intravenous analgesia.
  Interventions: Other: Standard intravenous analgesia.

INTERVENTIONS:
Procedure: BRILMA block — 20 ml 0.25 % bupivacaine was injected into the fascial plane between the serratus anterior muscle and the external intercostal muscle at T4 level.
  Arms: Group B: BRILMA block
Other: Standard intravenous analgesia. — Standard intravenous analgesia.
  Arms: Group C: Control

SUMMARY:
Regional analgesia technique in addition to multimodal analgesia in breast-conserving surgery aims to reduce opioid consumption. This study evaluates the postoperative analgesic efficacy of ultrasound-guided BRILMA block in patients undergoing breast conserving surgery.

DETAILED DESCRIPTION:
Breast-conserving surgery has become a standard surgical approach in the management of early-stage breast malignancies. Despite being less invasive than other oncologic procedures, postoperative pain remains a significant concern. In postoperative pain management, the addition of regional analgesia techniques to multimodal approaches aims to reduce opioid consumption.

First described in 2013, the Serratus-Intercostal Interfascial Plane block targets the branches of the intercostal nerves at the level of the mid-axillary line, specifically around the fourth rib-an anatomical region referred to by the acronym BRILMA. This regional anesthesia technique has demonstrated efficacy in managing postoperative pain, particularly after breast surgery.

In the study, investigators planned to evaluate the postoperative analgesic efficacy of ultrasound-guided BRILMA block via 24-hour morphine consumption in patients undergoing breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Breast-conserving surgery
* ASA I-III

Exclusion Criteria:

* Patient refusal
* Presence of contraindications for regional anesthesia ( bleeding disorder, infection at the injection site, local anesthetic allergy)
* Chronic analgesic use
* Preoperative breast pain
* BMI >35

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | postoperative 24-hour
  Amount of morphine consumption

SECONDARY OUTCOMES:
Static and dynamic pain scores assessed with numeric rating scale | postoperative 24 hours
  pain scores recorded at 0., 1., 4., 8., 12., 24. hours postoperatively
number of blocked dermatome | 20. minute after block performance
  pinprick test in mid-axillary and mid-claviculary line
Duration of block application | up to 15 minutes
  time from the insertion of probe to the removal of needle from skin
Amount of fentanyl for sedation. [Time Frame: Intraoperative 2-3 hours] | during surgery
  Amount fentanyl use during surgery
Rescue analgesia | postoperative 24 hours
  number of patients needed rescue analgesia
Nausea and vomit | postoperative 24 hours
  postoperative nausea and vomiting (0=no, 1= mild nausea, 2= severe nausea or vomiting)
Complications | Up to 24 hours
  Hematoma, vascular puncture, pneumothorax
Patient's satisfaction | Up to 24 hours
  Likert scale:1-5 (1: very dissatisfied, 5: very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Nükhet Sivrikoz, Assoc. Prof. Dr., Principal Investigator — Attending anesthesiologist
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)